CLINICAL TRIAL: NCT04789707
Title: Influence of Keratoconus on Stress at Work
Acronym: KERATOSTRESS
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2018 DUTHEIL 2; 2018-A02527-48 (Other: 2018-A02527-48)
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Keratoconus in One or Two Eyes for Case; Good Visual Acuity for Control
Keywords: keratoconus; Karasek; stress at work
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KERATOCONUS group: All workers with keratoconus all stages followed at the service of ophthalmology in CHU Gabriel Montpied, Clermont-Ferrand, Auvergne.
  The investigators only assessed data from usual routine practice. Patients answer the auto questionnaire in last minutes of consultation.
  Interventions: Behavioral: auto-questionnaire
- CONTROL group: workers with good visual acuity consulting in ophthalmology service of Clermont-Ferrand.
  The investigators only assessed data from usual routine practice. Patients answer the auto questionnaire in last minutes of consultation.
  Interventions: Behavioral: auto-questionnaire

INTERVENTIONS:
Behavioral: auto-questionnaire — Patients answer the auto questionnaire in last minutes of consultation.

SUMMARY:
Keratoconus is a progressive disorder in which central and paracentral corneal stromal thinning occurs.

No studies evaluated the influence of keratoconus on stress at work, nor the influence of treatments of keratoconus on stress at work, including Quality of Life at work and on perception of work. Moreover, it has been shown that some pathologies had greater influence in some occupations, also depending on other characteristics of individuals such as age, sex or socio professional groups.

Therefore, we hypothesized that keratoconus 1) will influence stress at work including QoL at work and perception of work, 2) will have a greater influence in some occupations and depending on age, sex, or stage of keratoconus, 3) will induce stoppage of work and occupational reclassifications.

DETAILED DESCRIPTION:
This is a descriptive, prospective, observational, monocentral study. For each patient with keratoconus and patient control, use of the auto questionnaire to carry out the study. we only assessed data from usual routine practice.

Stress at work is measured by Job Content Questionnaire of Karasek issued during consultations.

Study all workers the influence of keratoconus and its stage on:

* consequences of keratoconus in function of visual acuity, mode of correction and staging of the keratoconus.
* Psychological consequences: Quality of life at work, Perception of work (Karasek questionnaire), anxiety and depression (HAD scale)
* Professional consequences: stoppage of work and duration and occupational reclassifications
* Characteristics of the patient: age, sex, occupation.

Measures to reduce or avoid bias:

* Standardized, anonymous auto questionnaire
* A large workforce: high rate of participation is expected
* Inclusion of control group.

ELIGIBILITY:
Inclusion Criteria:

* patients with keratoconus all stages followed at the CHU Gabriel Montpied,
* patients constituting a representative control group of workers consulting in ophthalmology service of Clermont-Ferrand.

Exclusion Criteria:

* an other ophtalmological disease alters visual acuity.
* minors subjects
* inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with keratoconus patients constituting a representative control group of workers consulting in ophthalmology service of Clermont-Ferrand.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
stress at work | day 0
  measured by Job Content questionnaire of Karasek

SECONDARY OUTCOMES:
psychological consequences | Day 0
  measured by HAD scale
Stoppage of work | Day 0
  professional consequences of stoppage of work : reclassifications
Duration of stoppage of work | Day 0
  professional consequences of duration of stoppage of work : reclassifications
characteristics of the patient | day 0
  sex, age, occupation
Measure of visual acuity. | Day 0
  Consequence of keratoconous on visual acuity
Mode of correction. | Day 0
  visual consequences of keratoconus on mode of correction
staging of keratoconous | Day 0
  visual consequences of keratoconus on keratoconous stage

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU - Gabriel Montpied, Clermont-Ferrand, France